CLINICAL TRIAL: NCT03720587
Title: The Experiences of Patients With Greater Trochanteric Pain Syndrome.
Status: Completed | Type: Observational
Sponsor: The Royal Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ROH18ORTH15
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2018-10

CONDITIONS: Greater Trochanteric Pain Syndrome
Keywords: GTPS; Gluteal tendinopathy; Lateral hip pain; Trochanteric bursitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured interviews — Semi-struuctured telephone interviews

SUMMARY:
Greater Trochanteric Pain syndrome (GTPS) is a debilitating condition causing pain on the outside of the hip. This study aims to explore the experiences, beliefs and expectations of patients with GTPS, using semi-structured interviews.

DETAILED DESCRIPTION:
Greater Trochanteric Pain syndrome (GTPS) is a debilitating condition causing pain on the outside of the hip. There is growing evidence to suggest that psychological barriers to recovery are present in patients with peripheral pain. The experiences and beliefs of patients suffering with GTPS are unknown. This study aims to explore the experiences, beliefs and expectations of patients with GTPS, using semi-structured interviews to inform the development of interventions for evaluation in future research.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 16
* Able to speak and understand the English language
* Patients seen in a Specialist Consultant lead clinic who have been given the diagnosis of lateral hip pain, Greater Trochanteric Pain Syndrome (GTPS), Trochanteric Bursitis or Gluteal Tendinopathy.

Exclusion Criteria:

* Inflammatory conditions
* Systemic / Infective disease
* Previous diagnosis of Fibromyalgia or persistent multi-joint pain.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be identified from Orthopaedic clinic lists and the Outpatient Physiotherapy waiting list at a single, elective Orthopaedic NHS Trust. Patients will have been assessed in a Specialist Consultant lead clinic by and been given one of the following diagnoses:
  1. Lateral Hip pain
  2. Greater Trochanteric Pain Syndrome (GTPS)
  3. Trochanteric bursitis.
  4. Gluteal tendinopathy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Framework Method of data analysis. | 10 months
  A systematic approach to qualitative analysis specifically used when the objectives of a study are known, prior to analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Orthopaedic Hospital NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stephens G, O'Neill S, Mottershead C, Hawthorn C, Yeowell G, Littlewood C. "It's just like a needle going into my hip, basically all of the time". The experiences and perceptions of patients with Greater Trochanteric Pain syndrome in the UK National Health Service. Musculoskelet Sci Pract. 2020 Jun;47:102175. doi: 10.1016/j.msksp.2020.102175. Epub 2020 Apr 29. PMID 32452392